CLINICAL TRIAL: NCT06810518
Title: ALPCO Calprotectin CLIA Assay - Measurement of Calprotectin Levels in Human Stool
Status: Recruiting | Type: Observational
Sponsor: American Laboratory Products Company (Industry)
Responsible Party: Sponsor
Other Study IDs: ALPCO Calprotectin CLIA Study
Record Dates: First submitted 2025-01-31; First posted 2025-02-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis); Inflammatory Bowel Syndrome
Keywords: calprotectin; IBD; IBS
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- IBD: Adult subjects diagnosed with IBD via endoscopy and histological findings.
  Interventions: Device: ALPCO Calprotectin CLIA
- IBS: Adult subjects with IBS as per the Rome IV criteria.
  Interventions: Device: ALPCO Calprotectin CLIA
- Other GI Disorders: Adult subjects with gastrointestinal disorders not meeting the Rome IV criteria or IBD diagnosis.
  Interventions: Device: ALPCO Calprotectin CLIA
- Healthy Subjects: Adult subjects without any gastrointestinal complaints.
  Interventions: Device: ALPCO Calprotectin CLIA

INTERVENTIONS:
Device: ALPCO Calprotectin CLIA — Measurement of calprotectin in feces

SUMMARY:
The ALPCO Calprotectin CLIA is an in vitro diagnostic test intended to quantitatively measure concentrations of fecal calprotectin in human stool samples. Calprotectin is a protein biomarker of mucosal inflammation. Measurement of calprotectin can aid in the diagnosis of Inflammatory Bowel Diseases (IBD), specifically Crohn's Disease (CD) and Ulcerative Colitis (UC), as well as aid in the differentiation of IBD from Irritable Bowel Syndrome (IBS) when used in conjunction with other diagnostic testing and the total clinical picture. The goal of the study is to generate data to support positive and negative predictive value of the ALPCO Calprotectin assay in patients with signs and symptoms of IBS or IBD.

DETAILED DESCRIPTION:
The clinical study serves to confirm the sensitivity and specificity of the ALPCO Calprotectin CLIA as compared to gastroenterologist diagnosis (including colonoscopy results and other clinical information) in patients with signs and symptoms of IBS or IBD, using the proposed cut-off values (50 and 100 µg/g) as both an aid in the diagnosis of Inflammatory Bowel Disease and as an aid to differentiate IBD from Irritable Bowel Syndrome. The clinical study will be conducted in compliance with applicable requirements in the protection of human subjects regulations in 21 CFR part 50, the institutional review boards regulations in 21 CFR part 56, and the investigational device exemptions regulations in 21 CFR part 812.

The goal of this clinical study is to confirm the sensitivity and specificity of the ALPCO Calprotectin CLIA in patients using the proposed cut-off value (50 µg/g) as an aid in differentiating between a diagnosis of an Inflammatory Bowel Disease and other non-inflammatory disorders, most notably Irritable Bowel Syndrome. (See Appendix I for draft study protocol). Final assay cut-off will be determined upon completion of analytical studies and product validation.

Calprotectin values greater than 50 µg/g (or defined assay cut-off) are indicative of neutrophil infiltrate in the gastrointestinal tract, and therefore signal the presence of an active Inflammatory Bowel Disease. Calprotectin concentrations below this value do not indicate inflammation, but do not eliminate a potential diagnosis of Irritable Bowel Syndrome. Therefore, clinical use of the ALPCO Calprotectin CLIA can generate crucial data to determine whether or not a patient should undergo more invasive testing to diagnose the presence of an Inflammatory Bowel Disease. This clinical study will seek to confirm this conclusion by estimating the predictive value of positive and negative tests using the proposed cut off value in patients referred for diagnostic evaluation with signs and symptoms suggestive of either IBD or IBS.

The goal of the study is to generate data to support positive and negative predictive value of the ALPCO Calprotectin assay in patients with signs and symptoms of IBS or IBD.

This study will be performed at multiple clinical recruiting sites with a minimum of 3 analytical test sites - ALPCO would be one test site and could test all samples from collection sites only at which endoscopies (colonoscopy) focusing on the diagnosis of bowel inflammation are performed. Patients will be enrolled in the study based on inclusion/exclusion defined criteria.

All patients enrolled in the study with signs and symptoms of IBS or IBD, must provide a stool sample prior to having a scheduled endoscopy performed or shortly after the colonoscopy provided treatment has not begun and other inclusion/exclusion criteria have been met.

Patients enrolled in the study will be scheduled for a colonoscopy or would have had a colonoscopy in the timeframe listed in the inclusion criteria.

Results of the colonoscopy and histology will be used to determine disease status. Stool samples will be stored frozen until such time that they can be tested with the candidate device to determine the calprotectin measured value. Results of the ALPCO Calprotectin CLIA will be compared to the diagnosis obtained during the colonoscopy.

Agreement will be defined as follows:

A proposed cut-off of >50 µg/g Calprotectin represents a positive result indicating potential disease. A positive result must be confirmed by colonoscopy results indicating IBD. < 50 µg/g indicates a negative result.

Based on historical recruiting experience, approximately 220 or more patients with suspected IBD will be enrolled in the study with the goal of testing and enrolling

1. approximately 70 patients with a confirmed diagnosis of IBD (Crohn's Disease or Ulcerative Colitis);
2. approximately 100 patients with a confirmed diagnosis of Irritable Bowel Syndrome;
3. approximately 50 patients with IBD symptoms but a diagnosis of something other than IBD or IBS

All enrolled patients must meet the inclusion criteria for the appropriate study group and must provide a stool sample in accordance with protocol requirements. Additionally, we will recruit approximately 100 normal patients that will be tested only with the ALPCO Calprotectin CLIA. The normal patient groups will have no history of disease.

ELIGIBILITY:
Inclusion criteria:

* Male or female, ≥22 years of age (adults)
* Suspected inflammatory bowel disease or irritable bowel syndrome with symptoms such as abdominal pain, diarrhea, altered appetite, weight loss, or anemia
* Able to provide a sample according to the sampling protocol within 72-24 hours prior to the scheduled diagnostic endoscopy or 3-30 days after the colonoscopy.
* Able to understand the study and the tasks required and sign the ICF

Exclusion criteria:

* Unable or unwilling to provide a stool specimen
* Known active intestinal cancer or in remission with abnormal levels (per physician assessment)
* Known active intestinal infection or history of treated intestinal infection with persistent abnormal levels (per physician assessment)
* IBD patients receiving chemotherapy or systemic immunosuppressive drugs without completing an 8-week washout period
* IBD patients who have previously diagnosed IBD managed with immunomodulators, 5-ASA or biologic therapies without completing an 8-week washout period for biologics and immunomodulators or 4 weeks for 5-ASA
* IBD patients who have previously been diagnosed with IBD and have undergone a surgical resection or diversion procedure.
* Known upper Gl disease such as esophagitis or gastritis that might influence the study test's ability to detect intestinal inflammatory disease
* Have taken NSAIDS (including aspirin) on 7 or more days during the 2 weeks before providing the sample
* Samples are not collected according to sampling protocol.
* Any condition that in the opinion of the investigator should preclude participation in the study.

Using an IRB approved consent form, all study participants will be advised of study requirements and potential risks associated with study participation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals that presents with symptoms of IBS/IBD and otherwise healthy subjects
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
In vitro diagnostic value of Calprotectin | Through study completion, up to 52 weeks.
  Value of calprotectin measurement using the ALPCO Calprotectin CLIA on the chemiluminescent automated KleeYa instrument.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Med-Care Research Corp, Miami, Florida
  - ALPCO, Salem, New Hampshire
  - Gastro Intestinal Research Institute of Northern Ohio,, Westlake, Ohio

IPD SHARING:
Plan to Share IPD: No